CLINICAL TRIAL: NCT05844618
Title: A Randomized, Intraindividual, Phase 4 Study to Evaluate the Short-Term Efficacy of Triamcinolone Acetonide (Aristocort® C) in Subjects with Atopic Dermatitis
Brief Title: Short-Term Efficacy of Triamcinolone Acetonide (Aristocort® C) in Subjects with Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Inno-5011
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; aristocort; triamcinolone acetonide
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Intra-individual
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triamcinolone Acetonide (Aristocort® C) (Active Comparator)
  Interventions: Drug: Triamcinolone Acetonide (Aristocort® C)
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Triamcinolone Acetonide (Aristocort® C) — On Day 1, Day 2, and Day 3, subjects will receive 2 applications of 3 mg/cm2 on the same lesional area, at an interval of approximately 12 ± 2 hours.
  Arms: Triamcinolone Acetonide (Aristocort® C)
Drug: Vehicle — On Day 1, Day 2, and Day 3, subjects will receive 2 applications of 3 mg/cm2 on the same lesional area, at an interval of approximately 12 ± 2 hours.
  Arms: Vehicle

SUMMARY:
This study is a randomized, intraindividual study to evaluate the short-term efficacy of triamcinolone acetonide (Aristocort® C) in subjects with atopic dermatitis.

DETAILED DESCRIPTION:
This study is being conducted to evaluate the short-term efficacy and effect of triamcinolone acetonide (Aristocort® C) on pruritus, skin biomarkers and skin parameters in subject with atopic dermatitis.

Approximately 20 subjects with atopic dermatitis will receive twice-daily topical application of triamcinolone acetonide (Aristocort® C) or vehicle in two different randomized areas for 3 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age or older at the time of consent.
2. Subject has clinically confirmed diagnosis of active AD, according to Hanifin and Rajka criteria.
3. Subject has at least a 6-month history of AD and had no significant flares in AD for at least 4 weeks before screening.
4. Subject has 2 applications areas (10 X 10 cm) with a lesional surface of at least 6 X 6 cm, preferably located on 2 distinct anatomical areas at Day 1.

Exclusion Criteria:

1. Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
2. Subject has clinically infected AD.
3. Subject has a Fitzpatrick's Skin Phototype ≥5.
4. Subject has a history of skin disease or presence of skin condition, other than AD, that would interfere with the study assessments in the opinion of the investigator.
5. Subject is known to have immune deficiency or is immunocompromised.
6. Subject has a history of cancer or lymphoproliferative disease within 5 years prior to Day 1.
7. Subject has any clinically significant medical condition that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results.
8. Subject has a known history of chronic infectious disease.
9. Subject has a known or suspected allergy to triamcinolone acetonide (Aristocort® C) or any component of the investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pruritus NRS on AD lesions | 72 hours
  The intensity of pruritus will be evaluated using a NRS by asking subjects to assign a numerical score to the worst level of itching at each application area in the past 12 hours, on a scale from 0 to 10, where 0 indicates no itch and 10 indicates the worst imaginable itch.

SECONDARY OUTCOMES:
Change from baseline in pruritus NRS on AD lesions | 12, 24, 36, 48, and 60 hours
  The intensity of pruritus will be evaluated using a NRS (Numeric Rating Scale) by asking subjects to assign a numerical score to the worst level of itching at each application area in the past 12 hours, on a scale from 0 to 10, where 0 indicates no itch and 10 indicates the worst imaginable itch.
Change from baseline in skin biomarkers for AD | Day 2, Day 3, and Day 4
  An untargeted biomarker approach with gene expression profile of treated and untreated skin samples will be performed.
Change from baseline in TSS | Day 4
  The TSS (Total Sign Score) is an assessment of the severity of erythema, edema/papulation, oozing/crusting, excoriation, lichenification, and dryness, each scored independently using the 4-point severity scale with a value range from 0 to 3 (clear to severe). The rating for each parameter is then summed to create a score ranging from 0 to 18.
Change from baseline in TAA | Day 4
  The TAA (Target Areas Assessment) is a 6-point scale with a value range from 0 to 5 (clear to very severe) used to evaluate AD severity at each site of study drugs application.
Change from baseline in lesion IGA | Day 4
  The lesion IGA (Investigator Global Assessment) is a 5-point scale with a value range from 0 to 4 (clear to severe) used for the assessment of each target lesion severity.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (1):
- Innovaderm Research Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No